CLINICAL TRIAL: NCT06956625
Title: Cleansing Efficacy of Cosmetic Products - Particular Matter Model
Brief Title: Cleansing Efficacy of Cosmetic Product
Acronym: Cleanser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: SGS proderm GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 25.0054-60
Record Dates: First submitted 2025-04-23; First posted 2025-05-04 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Healthy Skin

STUDY DESIGN:
Intervention Model Description: Two test areas will be defined on both forearms. Area 1 will be located on the right forearm; Area 2 will be located on the left forearm. Treatments will be randomly and balanced assigned to the test areas.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cosmetic product (Experimental): Test area topically washed with cleanser containing Mitopure
  Interventions: Other: Topical cosmetic cleanser
- Tap water (control) (Other): Test area topically washed with tap water
  Interventions: Other: Topical tap water

INTERVENTIONS:
Other: Topical cosmetic cleanser — After applying the model pollutant, the test area will be topically cleaned with the active cosmetic cleanser with Mitopure.
  Arms: Cosmetic product
Other: Topical tap water — After applying the model pollutant, the test area will be topically cleaned with tap water (control).
  Arms: Tap water (control)

SUMMARY:
The aim of this study is to investigate the cleansing effect of one cosmetic product containing Mitopure against a particular matter model pollutant in comparison to an untreated control.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study
* Willingness to actively participate in the study and to come to the scheduled visits
* Female and/or male
* From 18 to 70 years of age
* Healthy skin in the test area
* Skin type on Fitzpatrick scale: I, II or III

Exclusion Criteria:

* Female subjects: Pregnancy or lactation
* Drug addicts, alcoholics
* AIDS, HIV-positive or infectious hepatitis
* Conditions which exclude a participation or might influence the test reaction/evaluation
* Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years
* Active skin disease at the test area
* Wounds, moles, tattoos, scars, irritated skin, excessive hair growth, etc. at the test area that could influence the investigation
* Any topical medication at the test area within the last 4 weeks prior to the start of the study and during the study
* Documented allergies to cosmetic products and/or ingredients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Luminosity (L) | Before pollutant application (t0), immediately after evaporation of the applied pollutant (t1), and 20 minutes after product rinse-off (t2)
  Luminosity in test area assessed by HiRIS (High Resolution Imaging System) image analysis will be used to quantify cleaning efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Katrin Unbereit, Principal Investigator — SGS proderm GmbH
Locations (1):
- SGS proderm GmbH, Schenefeld, Germany

IPD SHARING:
Plan to Share IPD: No